CLINICAL TRIAL: NCT04241900
Title: Effect of Aging and Aerobic Fitness Level on Heat Dissipation in Neutral Conditions
Brief Title: Effect of Aging and Aerobic Fitness Level on Heat Dissipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10. Aging and heat loss
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Risk of Heat Stress
Keywords: heat loss; aging; aerobic fitness level; heat stress
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shuttle run test (Experimental): At the shuttle run test, participants were required to run between two lines 20 meters apart, while keeping pace with audio signals emitted from a pre-recorded CD. The frequency of the sound signals increases in such way that running speed was increased by 0.5 km h-1 each minute from the starting speed 8.5 km h-1.
  Interventions: Behavioral: Shuttle run test

INTERVENTIONS:
Behavioral: Shuttle run test — At the shuttle run test, participants were required to run between two lines 20 meters apart, while keeping pace with audio signals emitted from a pre-recorded CD. The frequency of the sound signals increases in such way that running speed was increased by 0.5 km h-1 each minute from the starting speed 8.5 km h-1.

SUMMARY:
In the context of global aging, the health risk factors associated with exercising or working in the heat for aging population are exacerbated by the rising in global surface temperatures. The purpose of this investigation is to determine at what age the heat loss decrements occur and to examine if aerobic fitness level can affect the heat loss capacity in neutral environmental conditions.

DETAILED DESCRIPTION:
All trials were conducted to indoor gyms with the same environmental temperature and relative humidity, 26 - 30oC and 40-50% respectively, to ensure no difference in body temperature were due to the external thermal stress. The participants were instructed to refrain from intense exercise as well as alcohol and caffeine consumption for 24 hours prior to experimental trial and to had a light meal 2h before their arrival.

Upon arrival, participants would have to wear running shoes, light and short running shorts and light cotton socks. Participants received comprehensive instructions about the shuttle run test and the whole process of measurements. Firstly participants answered the International Physical Activity Questionnaire (IPAQ). Thereafter, anthropometrics data (weight and height) were evaluated as well as the body temperature in external ear canal and axillary. All participants followed five minutes warming up and then performed to 20 m shuttle run test until their volitional limit. Once the participants could no longer run, the test was over and the number of laps was recorded. After the end of the shuttle run, were evaluated the body temperature and the weight of each participants. No fluids consumptions were permitted until the second weighing. They were weighed twice, at baseline and at the end of the running test with a precision weight scale (Kern DE 150K2D, KERN & SOHN GmbH, Balingen, Germany).

Environmental data including air temperature and relative humidity were measured continuously using a portable weather station (LCD Digital Temperature & Humidity Meter HTC-1). The weather station was placed 1 meter above the ground according to the manufacturer's guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adults

Exclusion Criteria:

* Diagnosed chronic medical condition;
* Symptoms of acute illness;
* Recent (past 4 weeks) usage of medications known to affect the circulatory system, the thyroid, the pituitary function, or the metabolic status

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 431 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness level | Through study completion (a shuttle run test), an average of 15 minutes
  Aerobic fitness level was defined by peak oxygen uptake (VO2peak). VO2peak was determined by a 20m shuttle run test. The number of the last announced stage and the equivalent maximal speed from participants' performance were used for its VO2peak estimation
Change from baseline ear canal temperature | Change from baseline to the end of study completion (a shuttle run test), an average of 15 minutes
  Ear canal temperature was recorded twice, at baseline and at the end of the shuttle run test (three times each at the left ear and recorded the mean value), using ear thermometer (IR100, MicrolifeSwitzerland)
Change from baseline axillary temperature | Change from baseline to the end of study completion (a shuttle run test), an average of 15 minutes
  Axillary temperature was recorded twice, at baseline and at the end of the shuttle run test, using the electronic digital thermometer (EcoTemp, OMRON, Japan)
Physical activity levels | Once before the shuttle run test
  Physical activity of the subject in a usual week was recorded via International Physical Activity Questionnaire. Scores include steps/day and METs/week, with no lower and upper limit
Change from baseline body weight | Change from baseline to the end of study completion (a shuttle run test), an average of 15 minutes
  Weight was recorded twice, at baseline and at the end of the shuttle run test, using a precision weight scale (Kern DE 150K2D, KERN & SOHN GmbH, Balingen, Germany
Change from baseline whole Body Sweat Rate | Change from baseline to the end of study completion (a shuttle run test), an average of 15 minutes
  Whole Body Sweat Rate was determined by the difference of the pre-test and post-test weight of the participants
Air temperature | Up to 30 minutes, during a one complete shuttle run test
  Air temperature was measured continuously using a portable weather station (LCD Digital Temperature & Humidity Meter HTC-1placed) 1 meter above the ground according to the manufacturer's guidelines
Relative humidity | Up to 30 minutes, during a one complete shuttle run test
  Relative humidity was measured continuously using a portable weather station (LCD Digital Temperature & Humidity Meter HTC-1) placed 1 meter above the ground according to the manufacturer's guidelines

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Department of Exercise Science, University of Thessaly, Trikala, Thessaly
  - FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly

IPD SHARING:
Plan to Share IPD: Undecided